CLINICAL TRIAL: NCT05386992
Title: Anthropometric and Biomechanical Analysis of the Children's Foot for the Design of Healthy Footwear: ABIP Study
Brief Title: Anthropometric and Biomechanical Analysis of the Infant Foot
Acronym: ABIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABIP
Record Dates: First submitted 2022-05-15; First posted 2022-05-24 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Child, Only
Keywords: Children; Foot development; Foot posture; Paediatric foot; Shoes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anthropometric study of children's feet and healthy standard last design: (Experimental): An anthropometric study of the feet of the subjects included in the sample will be carried out. The variables of interest used in this work are collected by digitizing the foot and ankle of each person, as well as through an anonymous questionnaire, which the study volunteers and their parents or legal guardians fill out and deliver.
  From the data collected, 5 models of healthy standard last will be produced that are adapted to the anthropometric characteristics of our study population: sports last, boot last, sandal last, ballerina last and moccasin last.
  Interventions: Diagnostic Test: Anthropometric study

INTERVENTIONS:
Diagnostic Test: Anthropometric study — Once the 5 models of lasts have been produced in phase 1, certain shoe models will be designed and manufactured based on these lasts at random and at the free choice of the designers of a footwear company. These models will then be physically tested on children to analyze their effects on walking and walking.
  Other Names: Design and manufacture of shoes and fit tests

SUMMARY:
In the era of science and technology, footwear has become not only an essential item of clothing, but also another tool for the optimal development of children, the improvement of work and sports performance or the prevention and treatment of pathologies.

The anthropometric characteristics of the child's foot differ considerably from those of the adult foot, in fact, it is not until the age of 18-19 years that the structure of the foot is finally consolidated. Therefore, it is essential that footwear manufacturers know these characteristics to achieve an adequate design.

Current scientific evidence highlights the importance of considering the unique morphology of the infant foot, as well as the high functional demands to which footwear is subjected at these ages. There is a lack of studies that analyze in detail the shape of the child's foot.

DETAILED DESCRIPTION:
Given that the data we have so far comes from studies that are not very current and on small samples, there is a need to update these variables to transfer these results to the productive fabric.

Therefore, the objective of this research is to carry out an anthropometric and biomechanical analysis of the infant foot in order to use these data in the creation of a standard last that respects its morphology.

Subsequently, said last will be subjected to different fit tests to verify its correct adaptation to the foot in this population group.

ELIGIBILITY:
Inclusion Criteria:

* School-age boys and girls with foot sizes between 20 and 41
* Attending school and belonging to public, private or concerted schools, to guarantee the variability of the sample in terms of type of school.

Exclusion Criteria:

* Present a severe structural or functional alteration of the foot, which prevents an adequate digitization of the foot and ankle with the hardware and software used to collect the samples.
* Not having the signature of the informed consent or express authorization of the parents or legal guardians to carry out the measurement and the subsequent processing of the data.
* Inability to stand or walk independently.
* Present crying or fear, not being cooperative or engaging in inappropriate behavior.

Ages: 12 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1216 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
Shoe test | Up to 3 month
  Using different reference points of the foot, the areas to be measured will be measured in millimeters. They are collected by digitizing the foot and ankle of each person, using the 3D scanner and the IcadPie Software.
Plantar pressure | Up to 3 month
  Based on sensory technology, the sensors are placed along a fixed platform, connected via a universal serial bus cable to a computer and appropriate software. The sensors, by supporting pressure, generate a potential difference that can be measured. This electrical voltage value is detected by the sensors themselves, and a computer program reinterprets it in the form of a graph with the captured values. The graph consists of a plantar footprint with a range of colors, according to the relative baropressure captured.
  This instrument would provide us with quantifiable data about how load patterns behave in bare feet and shoes, in order to establish useful comparisons in our study

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez Suárez, PhD, Study Chair — University of Las Palmas de Gran Canaria
Locations (1):
- Manuel Pereira Domínguez., Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez C, De Vera M, Chhina H, Black A. Normative data for the dynamic pedobarographic profiles of children. Gait Posture. 2008 Aug;28(2):309-15. doi: 10.1016/j.gaitpost.2008.01.017. Epub 2008 Apr 15. PMID 18417345
- [Result] Beulertz J, Bloch W, Prokop A, Rustler V, Fitzen C, Herich L, Streckmann F, Baumann FT. Limitations in Ankle Dorsiflexion Range of Motion, Gait, and Walking Efficiency in Childhood Cancer Survivors. Cancer Nurs. 2016 Mar-Apr;39(2):117-24. doi: 10.1097/NCC.0000000000000256. PMID 25881810
- [Result] Bok SK, Lee H, Kim BO, Ahn S, Song Y, Park I. The Effect of Different Foot Orthosis Inverted Angles on Plantar Pressure in Children with Flexible Flatfeet. PLoS One. 2016 Jul 26;11(7):e0159831. doi: 10.1371/journal.pone.0159831. eCollection 2016. PMID 27458719
- [Result] Buckland MA, Slevin CM, Hafer JF, Choate C, Kraszewski AP; Hospital for Special Surgery Pediatric Research Team. The effect of torsional shoe flexibility on gait and stability in children learning to walk. Pediatr Phys Ther. 2014 Winter;26(4):411-7. doi: 10.1097/PEP.0000000000000084. PMID 25251796
- [Result] Gonzalez Elena ML, Cordoba-Fernandez A. Footwear fit in schoolchildren of southern Spain: a population study. BMC Musculoskelet Disord. 2019 May 10;20(1):208. doi: 10.1186/s12891-019-2591-3. PMID 31077163
- [Derived] Dominguez MP, Blanco SG, Paralera-Morales C, Martinez AR, Quintana-Montesdeoca MP, Baez-Suarez A. Anthropometric Foot Variations in Children: A Cross-Sectional Study Supporting Sex-Based Last Design. J Foot Ankle Res. 2025 Sep;18(3):e70069. doi: 10.1002/jfa2.70069. PMID 40746028